CLINICAL TRIAL: NCT02030665
Title: Individualized Assessment and Treatment for Marijuana Dependence: Treatment Mechanisms
Brief Title: Marijuana Treatment Project 4
Acronym: MTP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 12-174-3; R01DA012728 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Marijuana Dependence
Keywords: Marijuana Dependence; Individualized treatment; Motivational Enhancement Treatment; Cognitive-Behavioral Treatment; Contingency Management
MeSH Terms: conditions — Marijuana Abuse | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standardized MET plus CB (SMET-CB) (Active Comparator): Motivational Enhancement plus Cognitive-Behavioral treatment
  Interventions: Behavioral: Cognitive-Behavioral Treatment
- SMET+ CM (SMET-CB-CM) (Experimental): Motivational Enhancement plus CB treatment plus contingency management
  Interventions: Behavioral: Contingency Management
- Individualized Assessment & Treatment (IATP) (Experimental): Individualized Assessment and Treatment Program; Cognitive-Behavioral Treatment based on in-depth field monitoring of patient behavior
  Interventions: Behavioral: Individualized Assessment & Treatment
- IATP + CM (IATP-CM). (Experimental): Individualized Assessment and Treatment plus Contingency Management
  Interventions: Behavioral: Contingency Management; Behavioral: Individualized Assessment & Treatment

INTERVENTIONS:
Behavioral: Contingency Management — Reinforcement provided contingent upon demonstration of negative drug tests
  Other Names: Positive Reinforcement
  Arms: IATP + CM (IATP-CM).; SMET+ CM (SMET-CB-CM)
Behavioral: Individualized Assessment & Treatment — Tailored Cognitive-Behavioral Treatment based on detailed records of patient behavior
  Other Names: IATP
  Arms: IATP + CM (IATP-CM).; Individualized Assessment & Treatment (IATP)
Behavioral: Cognitive-Behavioral Treatment — Standard psychoeducational approach to coping skills training
  Other Names: CBT
  Arms: Standardized MET plus CB (SMET-CB)

SUMMARY:
Marijuana is the most commonly used illicit drug in the US, but treatment for marijuana dependence is not fully effective. In the current proposal we are exploring the idea that more tailored teaching of coping skills may result in improved outcomes for marijuana-dependence than those seen thus far. Participants will be 275 men and women meeting criteria for marijuana dependence and randomly assigned to 9 sessions of treatment in one of 4 treatment conditions: Standardized MET plus CB (SMET-CB); SMET+ CM (SMET-CB-CM); IATP; or IATP + CM (IATP-CM). Patients in all treatments will engage in ES via cell-phone for two weeks prior to treatment, for a weekly period during treatment, for another week after treatment has ended, and for two weekly periods at months 8 and 14. In the IATP conditions, the information gathered from the pretreatment and during-treatment ES periods will provide data for a functional analysis of patients' drug use and urges to use. It is hypothesized that IATP conditions will yield significantly better coping skills acquisition than SMET-CB conditions, both at posttreatment and at extended follow-ups, and that change in coping skills will predict better outcomes for the IATP conditions

DETAILED DESCRIPTION:
Marijuana is the most commonly used illicit drug in the US, but treatment for marijuana dependence is not fully effective. The most effective treatments to date have employed motivational enhancement (MET) plus cognitive-behavioral coping skills treatment (CB) and contingency management (CM) for abstinence. This proposal is a competitive renewal of our recently completed study to enhance coping and self-efficacy to improve marijuana outcomes in the long term. In the current proposal we are exploring the idea that more tailored teaching of coping skills may result in improved outcomes for marijuana-dependence than those seen thus far. The Individualized Assessment and Treatment Program (IATP) for marijuana dependent patients will employ experience sampling (ES) to determine the strengths and weaknesses of each patient in drug-use situations so that treatment can be tailored accordingly. Results from a pilot study indicated that IATP for alcohol dependent patients yielded better drinking outcomes at posttreatment than a packaged CB program (PCBT), that IATP patients reported greater use of coping skills than PCBT participants, and that posttreatment reports of coping skills were related to posttreatment drinking. Participants will be 275 men and women meeting criteria for marijuana dependence and randomly assigned to 9 sessions of treatment in one of 4 treatment conditions: Standardized MET plus CB (SMET-CB); SMET+ CM (SMET-CB-CM); IATP; or IATP + CM (IATP-CM). Patients in all treatments will engage in ES via cell-phone for two weeks prior to treatment, for a weekly period during treatment, for another week after treatment has ended, and for two weekly periods at months 8 and 14. In the IATP conditions, the information gathered from the pretreatment and during-treatment ES periods will provide data for a functional analysis of patients' drug use and urges to use. Therapists will use the information to address specific cognitions, affects, and behaviors that are adaptive and maladaptive, and will tailor a specific coping skills program with the patient. During-treatment experience sampling will allow adjustment of the treatment goals and procedures, making the treatment adaptive. In the SMET-CB conditions the experience sampling data will not be used in therapy, but will still provide in-vivo measures of drinking and coping skills. It is hypothesized that IATP conditions will yield significantly better coping skills acquisition than SMET-CB conditions, both at posttreatment and at extended follow-ups, and that change in coping skills will predict better outcomes for the IATP conditions. It is further predicted that the addition of CM to both IATP and SMET-CB will enhance short-term and long-term outcomes. The results will have implications for improved tailoring of treatment to patients' strength and deficits, and for the validity of the training of coping skills for relapse prevention. The data collected will shed light on the ways in which patients in treatment use coping skills in real-time contexts. Finally, the use of repeated ES periods will allow us to determine how treatment impacts thoughts, feelings and behaviors, and how these in turn affect outcome in the long and short term.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 yrs old
* meet Diagnostic and Statistical Manual IV (DSM-IV) criteria for Cannabis Dependence
* be willing to accept random assignment to any of the 4 treatment conditions

Exclusion Criteria:

* acute medical/psychiatric problems that require inpatient treatment (e.g., acute psychosis, severe depression, suicide/homicide risk)
* reading ability below the fifth grade level
* lack of reliable transportation
* excessive commuting distance.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Marijuana Use | every 3 months
  Marijuana use measured in terms of Days of use in every 90-day period

SECONDARY OUTCOMES:
Coping Skills | every 3 months
  Coping Skills measured using the Coping Skills Survey, administered every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, PhD, Principal Investigator — UConn Health; Elise Kabela-Cormier, PhD, Study Director — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Litt MD, Kadden RM, Tennen H, Dunn HK. Momentary coping and marijuana use in treated adults: Exploring mechanisms of treatment. J Consult Clin Psychol. 2021 Apr;89(4):264-276. doi: 10.1037/ccp0000633. PMID 34014689
- [Derived] Litt MD, Kadden RM, Tennen H, Petry NM. Individualized assessment and treatment program (IATP) for cannabis use disorder: Randomized controlled trial with and without contingency management. Psychol Addict Behav. 2020 Feb;34(1):40-51. doi: 10.1037/adb0000491. Epub 2019 Jul 18. PMID 31318225